CLINICAL TRIAL: NCT01698307
Title: A Cluster Randomized Controlled Trial of an Enhanced Treatment Algorithm for the Management of Crohn's Disease
Brief Title: Enhanced Algorithm for Crohn's Treatment Incorporating Early Combination Therapy
Acronym: REACT2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alimentiv Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP1202
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Deep Remission; Complications
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

STUDY DESIGN:
Intervention Model Description: algorithm
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Treatment Algorithm (Active Comparator): The Enhanced algorithm features the early use of combined antimetabolite/adalimumab therapy, and treatment intensification based on ileocolonoscopic findings. Failure to achieve or sustain Deep Remission, which includes sustained normalization of the imaging studies, will result in treatment intensification, according to the steps outlined in the algorithm, irrespective of symptoms.
  Interventions: Other: Enhanced Treatment Algorithm
- Conventional Step-care Algorithm (Other): Step-care algorithm that specifies treatment escalation solely on the basis of symptoms quantified using the Harvey Bradshaw Index (HBI).
  Interventions: Other: Conventional Step-care Algorithm

INTERVENTIONS:
Other: Enhanced Treatment Algorithm — The Enhanced algorithm features the early use of combined antimetabolite/adalimumab therapy, and treatment intensification based on ileocolonoscopic findings. Failure to achieve or sustain Deep Remission, which includes sustained normalization of the imaging studies, will result in treatment intensification, according to the steps outlined in the algorithm, irrespective of symptoms.
  Other Names: Adalimumab
  Arms: Enhanced Treatment Algorithm
Other: Conventional Step-care Algorithm — Step-care algorithm that specifies treatment escalation solely on the basis of symptoms quantified using the Harvey Bradshaw Score.
  Arms: Conventional Step-care Algorithm

SUMMARY:
Assess if the implementation of an enhanced treatment algorithm will improve the management Crohn's Disease compared to a conventional Step-care approach.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a chronic inflammatory disorder of the gastrointestinal tract. During disease exacerbations, pharmacological or surgical intervention is usually needed to re-establish remission. Ideally, strategies should be employed to maintain patients in long-term remission while minimizing exposure to corticosteroids and reduce therapy-related toxicity.

Nevertheless, in reality many patients with CD do not receive effective therapy and their disease often remains active, leading to uncontrolled inflammation and complications from either the underlying disease or corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of CD
* Written informed consent must be obtained and documented.
* Willing to utilize study supply of adalimumab provided in syringe format, if indicated according to treatment algorithm.

Exclusion Criteria:

* Any conditions (e.g., history of alcohol or substance abuse) which, in the opinion of the investigator, may interfere with the patient's ability to comply with study procedures.
* Latex allergy or other conditions in which adalimumab syringes are contraindicated
* Currently participating, or planning to participate in a study involving investigational product within 24 months that may interfere with the patient's ability to comply with study procedures.
* Previously failed all classes of tumor necrosis factor (TNF) antagonists for the treatment of CD.
* Diagnosis of short bowel syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1095 (Actual)
Dates: Start 2014-03-28 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
Risk of Crohn's Disease-related complications at two years | 2 years
  Crohn''s Disease (CD)-related complications include (1) CD-related surgeries and non-surgical CD events (such as disease flare, bowel obstruction, and bowel damage events (such as symptomatic bowel obstruction, fistula, abscess and CD related hospitalizations and 2) complications and hospitalizations related to CD medications or procedures.

SECONDARY OUTCOMES:
Risk of Crohn's Disease-related complications, Crohn's Disease-related hospitalizations, and all cause hospitalizations at 6 months and 12 months. | six months, 12 months
  Crohn's Disease (CD)-related complications include (1) CD-related surgeries and non-surgical CD events (such as disease flare, bowel obstruction, and bowel damage events (such as symptomatic bowel obstruction, fistula, abscess and CD related hospitalizations and 2) complications and hospitalizations related to CD medications or procedures.
Time to first Crohn's Disease-related complication, first Crohn's Disease-related hospitalizations, and first all cause hospitalizations at 6 months and 12 months. | six months, 12 months
  Crohn's Disease (CD)-related complications include (1) CD-related surgeries and non-surgical CD events (such as disease flare, bowel obstruction, and bowel damage events (such as symptomatic bowel obstruction, fistula, abscess and CD related hospitalizations and 2) complications and hospitalizations related to CD medications or procedures.

OTHER OUTCOMES:
Proportion of patients at one year and two years who are in Deep Remission without disease progression | 1 year, 2 years
  Disease progression is defined as the de novo development of strictures or fistula, the occurrence of an intra-abdominal abscess, or surgery for Crohn's Disease (resection, bypass, stricturoplasty).
Proportion of patients at one year and two years who are in Deep Remission | 1 year, 2 years
  Deep remission defined as a Harvey-Bradshaw Index (HBI) less than or equal to 4, no steriods for the treatment of Crohn's Disease, and normal C-reactive protein
Proportion of patients at one year and 2 years who are in Clinical Remission | 1 year, 2 years
  Clinical remission defined as an Harvey-Bradshaw Index (HBI) of equal to or less than 4.
Change in C-reactive protein | 6 months, 1 year, 2 years
Change in health related QoL, patient and physician global rating | 6 months, 1 year, 2 years
  The EuroQoL instrument [EQ-5D] will be used to measure quality of life.
Patient and physician satisfaction | 2 years
  At the completion of study participation, subjects and physicians in both treatment groups will be asked to complete a satisfaction questionnaire regarding the information provided and their overall satisfaction with the approach to the management of CD. The physicians will also be asked if they would recommend the CD treatment algorithm to their colleagues, and if they think it would be feasible to sustain this algorithm within their practice setting.

CONTACTS AND LOCATIONS:
Overall Officials: Brian G Feagan, MD, Principal Investigator — Robarts Clinical Trials - Western University
Locations (22):
- United States (5):
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Carle Foundation Hospital, Urbana, Illinois
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Asheville Gastroenterology Associates, PA, Asheville, North Carolina
  - Scott and White Memorial Hospital, Temple, Texas
- Canada (7):
  - Duane Sheppard, GI Inc., Dartmouth, Nova Scotia
  - The Office of Dr. Bruce Musgrave, Kentville, Nova Scotia
  - Dr. Fashir Medical Inc., Sydney, Nova Scotia
  - Sudbury Endoscopy Center, Greater Sudbury, Ontario
  - S. and T. Shulman Medicine Professional Corporation, North Bay, Ontario
  - Oravec Medicine Professional Corporation, Oshawa, Ontario
  - The Office of Dr. Pierre Laflamme, Saint-Charles-Borromée, Quebec
- Germany (3):
  - Verein fur Wissenschaft und Fortbildung, Oldenburg, Lower Saxony
  - Praxis fur Gastroenterologie am Bayerischen Platz, Berlin
  - Gastroenterologie Eppendorfer Baum, Hamburg
- United Kingdom (7):
  - Royal Berkshire NHS Foundation Trust, Reading, Berkshire
  - The Royal Bournemouth Hospital, Bournemouth, Dorset
  - The Royal Hampshire County Hospital, Winchester, Hampshire
  - Oxford University Hospitals NHS Foundation - John Radcliffe Hospital, Headington, Oxford
  - University Hospital Coventry, Coventry, West Midlands
  - New Cross Hospital - Royal Wolverhampton NHS Trust, Wolverhampton, West Midlands
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: No
The study is site randomization not subject.

REFERENCES:
- [Background] Colombel JF, Rutgeerts PJ, Sandborn WJ, Yang M, Camez A, Pollack PF, Thakkar RB, Robinson AM, Chen N, Mulani PM, Chao J. Adalimumab induces deep remission in patients with Crohn's disease. Clin Gastroenterol Hepatol. 2014 Mar;12(3):414-22.e5. doi: 10.1016/j.cgh.2013.06.019. Epub 2013 Jul 12. PMID 23856361
- [Background] Feagan BG, Panaccione R, Sandborn WJ, D'Haens GR, Schreiber S, Rutgeerts PJ, Loftus EV Jr, Lomax KG, Yu AP, Wu EQ, Chao J, Mulani P. Effects of adalimumab therapy on incidence of hospitalization and surgery in Crohn's disease: results from the CHARM study. Gastroenterology. 2008 Nov;135(5):1493-9. doi: 10.1053/j.gastro.2008.07.069. Epub 2008 Aug 3. PMID 18848553
- [Background] Colombel JF, Sandborn WJ, Reinisch W, Mantzaris GJ, Kornbluth A, Rachmilewitz D, Lichtiger S, D'Haens G, Diamond RH, Broussard DL, Tang KL, van der Woude CJ, Rutgeerts P; SONIC Study Group. Infliximab, azathioprine, or combination therapy for Crohn's disease. N Engl J Med. 2010 Apr 15;362(15):1383-95. doi: 10.1056/NEJMoa0904492. PMID 20393175
- [Background] D'Haens G, Baert F, van Assche G, Caenepeel P, Vergauwe P, Tuynman H, De Vos M, van Deventer S, Stitt L, Donner A, Vermeire S, Van De Mierop FJ, Coche JR, van der Woude J, Ochsenkuhn T, van Bodegraven AA, Van Hootegem PP, Lambrecht GL, Mana F, Rutgeerts P, Feagan BG, Hommes D; Belgian Inflammatory Bowel Disease Research Group; North-Holland Gut Club. Early combined immunosuppression or conventional management in patients with newly diagnosed Crohn's disease: an open randomised trial. Lancet. 2008 Feb 23;371(9613):660-667. doi: 10.1016/S0140-6736(08)60304-9. PMID 18295023
- [Background] Lichtenstein GR, Feagan BG, Cohen RD, Salzberg BA, Diamond RH, Chen DM, Pritchard ML, Sandborn WJ. Serious infections and mortality in association with therapies for Crohn's disease: TREAT registry. Clin Gastroenterol Hepatol. 2006 May;4(5):621-30. doi: 10.1016/j.cgh.2006.03.002. PMID 16678077
- [Derived] Ungaro RC, Colombel JF. Treat to target with ustekinumab for Crohn's disease. Lancet Gastroenterol Hepatol. 2022 Apr;7(4):276-277. doi: 10.1016/S2468-1253(22)00019-X. Epub 2022 Feb 1. No abstract available. PMID 35120657